CLINICAL TRIAL: NCT02944123
Title: An Open-label, Randomized, Prospective Study Exploring Half Dose of Prasugrel and Ticagrelor in Platelet Response After Acute Coronary Syndromes
Brief Title: Half Dose of Prasugrel and Ticagrelor in Acute Coronary Syndrome (HOPE-TAILOR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Moo Hyun Kim, Professor, Dept. of Cardiology Dong-A University Hospital, Dong-A University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HOPE-TAILOR
Record Dates: First submitted 2016-10-24; First posted 2016-10-25 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Acute Coronary Syndrome
Keywords: Half dose; Newer oral P2Y12 receptor inhibitors; Acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel; Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Open-labeled
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Clopidogrel 75 mg (Other): Clopidogrel 600 mg as loading dose and followed by 75 mg/day as maintenance dose.
  Interventions: Drug: Clopidogrel 75 mg
- Prasugrel 5 mg (Experimental): Loading / maintenance dose: prasugrel 60 mg / 10 mg/day; After 1-month treatment of conventional dose, followed half dose of 5 mg/day for chronic treatment.
  Interventions: Drug: Prasugrel 5 mg
- Ticagrelor 45 mg (Experimental): Loading / maintenance dose: ticagrelor 180 mg / 90 mg/bid; After 1-month treatment of conventional dose, followed half dose of 45 mg/bid for chronic treatment.
  Interventions: Drug: Ticagrelor 45 mg

INTERVENTIONS:
Drug: Clopidogrel 75 mg — Clopidogrel 600 mg as loading dose followed by 75 mg/day as maintenance dose.
  Other Names: Plavix 75 mg
  Arms: Clopidogrel 75 mg
Drug: Prasugrel 5 mg — Loading / maintenance dose: prasugrel 60 mg / 10 mg/day; After 1-month treatment of conventional dose, followed half dose of 5 mg/day for chronic treatment.
  Other Names: Effient 5 mg
  Arms: Prasugrel 5 mg
Drug: Ticagrelor 45 mg — Loading / maintenance dose: ticagrelor 180 mg / 90 mg/bid; After 1-month treatment of conventional dose, followed half dose of 45 mg/bid for chronic treatment.
  Other Names: Brilinta 45 mg
  Arms: Ticagrelor 45 mg

SUMMARY:
East Asian patients will be required optimal dose of newer P2Y12 inhibitors (prasugrel or ticagrelor) to determine the safer treatment and better outcome. Whether lower dose of these regimens are more adequate for clinical practice in Korea is unclear. Therefore, the investigators aim to evaluate efficacy and safety of half dose of new oral P2Y12 inhibitors in Korean patients with acute coronary syndrome (ACS) undergoing percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
In recent years, newer oral P2Y12 receptor blockers (prasugrel or ticagrelor) have been strong recommendations for management of patients with ACS undergoing (PCI). These drugs provided more profound inhibitory effects than clopidogrel, which could lead to marked reduction in ischemic events, with relatively increase in bleeding complication, specific to low body weight, especially in women and East Asian patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients present with acute coronary syndrome undergoing primary PCI.
* Patients receive DAPT (conventional dose of P2Y12 inhibitors+aspirin) at least 1 month.
* Patients provide written informed consent prior to enrollment.

Exclusion Criteria:

* Low body weight (<60kg).
* History of transient ischemic attack or stroke.
* History of upper gastrointestinal bleeding in recent 6 months.
* Renal dysfunction defined as serum creatinine > 2.5 mg/dl
* Severe hepatic dysfunction defined as serum transaminase > 3 times normal limit
* On treatment with oral anticoagulant (Vitamin K antagonists, dabigatran, rivaroxaban).
* Bleeding tendency.
* Thrombocytopenia defined by platelet < 100,000/ml.
* Anemia defined by hemoglobin < 10 g/dl.
* Current treatment with drugs interfering with CYP3A4 metabolism (to avoid interaction with Ticagrelor): Ketoconazole, itraconazole, voriconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, and telithromycin.
* Known severe chronic obstructive pulmonary disease or bradycardia (sick sinus syndrome (SSS) or high degree AV block without pacemaker protection).
* Contraindication for study drugs.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Optimal platelet reactivity (OPR) rate | At post-PCI 3 months.
  OPR, indicate 85 to 208 for P2Y12 reaction units (PRU) or 16% to 50% for vasodilator-stimulated phosphoprotein (VASP)-platelet reactivity index (PRI)

SECONDARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCE) | Post-PCI 6 months.
  MACCE: composite of cardiac death, non-fatal myocardial infarction, repeat revascularization and stroke
Bleeding events | Post-PCI 6 months.
  BARC: Bleeding Academic Research Consortium (BARC ≥2).
Drug side effects | Post-PCI 6 months.
  Dyspnea or ventricular pauses ≥3 sec

CONTACTS AND LOCATIONS:
Overall Officials: Moo Hyun Kim, MD, Principal Investigator — Dong-A University Hospital
Locations (1):
- Dong-A University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goto S, Huang CH, Park SJ, Emanuelsson H, Kimura T. Ticagrelor vs. clopidogrel in Japanese, Korean and Taiwanese patients with acute coronary syndrome -- randomized, double-blind, phase III PHILO study. Circ J. 2015;79(11):2452-60. doi: 10.1253/circj.CJ-15-0112. Epub 2015 Sep 16. PMID 26376600